CLINICAL TRIAL: NCT05723588
Title: Neuroimaging Correlates and Feasibility of Transcranial Magnetic Stimulation (TMS) to Improve Smoking Cessation Outcomes in Veterans With Comorbid PTSD
Acronym: TMS-STOP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NURA-001-22S; 1625460 (Other: VA IRBNet identifier); CX002610 (Other Grant/Funding Number: eRA)
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco use cessation; Veterans
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation | interventions — Cognitive Behavioral Therapy; Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will receive either active repetitive transcranial magnetic stimulation (rTMS) or sham rTMS. Participants and the PI, who provides the rTMS will be blinded to this condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active rTMS (Experimental): Participants assigned to this group will receive active repetitive transcranial magnetic stimulation (rTMS) as part of their smoking cessation treatment.
  Interventions: Device: active repetitive transcranial magnetic stimulation; Behavioral: cognitive behavioral therapy for smoking cessation; Drug: nicotine replacement therapy
- sham rTMS (Sham Comparator): Participants assigned to this group will receive sham repetitive transcranial magnetic stimulation (rTMS) as part of their smoking cessation treatment.
  Interventions: Device: sham repetitive transcranial magnetic stimulation; Behavioral: cognitive behavioral therapy for smoking cessation; Drug: nicotine replacement therapy

INTERVENTIONS:
Device: active repetitive transcranial magnetic stimulation — Active rTMS is a non-invasive brain stimulation intervention that is FDA cleared as a treatment for smoking cessation in adults.
  Other Names: active rTMS
  Arms: active rTMS
Device: sham repetitive transcranial magnetic stimulation — Sham rTMS involves no brain stimulation, but appears to the participant and provider to be active rTMS.
  Other Names: sham rTMS
  Arms: sham rTMS
Behavioral: cognitive behavioral therapy for smoking cessation — All participants will receive five sessions of cognitive behavioral therapy (CBT) for smoking cessation.
  Other Names: CBT
Drug: nicotine replacement therapy — All participants will receive nicotine replacement therapy in for the form of 21 mg, 14 mg, and/or 7 mg nicotine patches (based on smoking quantity) and a "rescue" method such as nicotine lozenge or nicotine gum.
  Other Names: NRT, nicotine patch, nicotine gum, nicotine lozenges

SUMMARY:
Tobacco use is the number one preventable cause of the death in the United States, and is high among US Veterans, and those who have experienced trauma are more likely to smoke. Despite the efficacy of current evidence-based treatments for smoking cessation, there is a critical need for alternative treatments. This project seeks to evaluate the feasibility and effectiveness of a smoking cessation treatment for Veterans with posttraumatic stress disorder (PTSD) who smoke. The treatment combines smoking cessation counseling, nicotine replacement therapy (e.g., nicotine gum), and repetitive transcranial magnetic stimulation (rTMS). rTMS is a noninvasive brain stimulation treatment that has been cleared by the Food and Drug Administration for smoking cessation in adults.

DETAILED DESCRIPTION:
Tobacco use remains the number one preventable cause of death in the United States. Unfortunately, individuals with mental health conditions are disproportionately affected. Tobacco use is also high among US Veterans, and those who have experienced trauma are even more likely to smoke. Successful quitting is especially difficult for individuals who develop posttraumatic stress disorder (PTSD). Despite the efficacy of current evidence-based pharmacotherapies and psychotherapies for smoking cessation, alternative treatments are critically needed. Neuroimaging techniques such as resting-state functional magnetic resonance imaging (rs-fMRI) have provided insight into the neurocircuitry of tobacco use disorder (TUD) and successful quit attempts. Interventions that modulate the neural systems underlying TUD, such as repetitive transcranial magnetic stimulation (rTMS), may be critical to improving clinical outcomes. Indeed, the US Food and Drug Administration (FDA) recently cleared a form of rTMS as a short-term smoking cessation treatment in adults. However, most clinical trials on rTMS for smoking cessation have been conducted in civilian samples and have excluded individuals with psychiatric conditions. To improve smoking cessation treatment options for Veterans with PTSD, it is critical to evaluate novel brain stimulation methods such as rTMS in this vulnerable population. Furthermore, the development of neuroscience-informed techniques to enhance rTMS such as neuronavigation based on rs-fMRI is critical to individualizing rTMS for smoking cessation and understanding mechanisms of action. The application of neuroimaging to develop personalized rTMS targets to precisely modulate targeted underlying neurocircuitry has been successfully applied to the treatment of major depressive disorder (MDD). Similar methodology has been demonstrated successfully for smoking cessation by the candidate's mentors, but this work was completed in a sample of civilian participants making a quit attempt who did not have psychiatric illness. To fill these knowledge gaps, the proposed research aims to develop feasibility data for the therapeutic application individualized neuronavigated rTMS for Veterans with PTSD attempting to quit smoking. Using a feasibility randomized controlled trial (RCT) design, eligible Veterans with PTSD (n=50) seeking smoking cessation will receive rs-fMRI before and after a 5-day course of neuronavigated rTMS the week prior to their quit date, in conjunction with nicotine replacement therapy (NRT) and cognitive behavioral therapy (CBT). The scientific aims of the study are to evaluate feasibility of treatment delivery procedures, develop preliminary effect size estimates, and demonstrate target engagement of the intervention within neural networks critical to TUD.

ELIGIBILITY:
Inclusion Criteria:

* Is a US Veteran
* Meets DSM-5 criteria for tobacco use disorder
* Is between the ages of 18 and 75
* Smokes an average of 10 cigarettes per day for the past 6 months, with carbon monoxide (CO) level > 6 ppm
* Is willing to attempt smoking cessation
* Meets DSM-5 criteria for current PTSD diagnosis
* Speaks, reads and writes English
* Is willing to sign a Duke consent for those portions of the study that occur at Duke
* Has been stable on psychotropic medications for at least three months

Exclusion Criteria:

* Has had a substance use disorder other than tobacco in the preceding 3 months
* Has a history of myocardial infarction in the past 6 months or has another contraindication to NRT
* Has a contraindication to TMS or MRI

  * Personal or family history of a seizures or epilepsy
  * History of neurological condition that increases the risk of seizures including stroke or transient ischemic attack, cerebral aneurysm, or severe traumatic brain injury from a penetrating head injury, loss of consciousness > 20 minutes at time of traumatic injury, requiring an anticonvulsant medication for seizures, and/or found to have encephalomalacia on baseline MRI
  * Structural brain lesion, or prior brain surgery
  * Ferromagnetic metal in head (including shrapnel)
  * Implanted devices that may be affected by MRI or TMS (pacemaker, medication pump, cochlear implant, implanted deep brain stimulator)
  * Is pregnant (to be determined at Duke)
* Is unable to complete study procedures
* Is currently prescribed bupropion and/or varenicline
* Uses other forms of nicotine such as cigars, pipes, chewing tobacco, or vaping
* Is unable to provide informed consent due to a major neurocognitive disorder or other reason
* Meets criteria for a primary psychotic disorder or current manic episode
* Is currently imprisoned or psychiatrically hospitalized
* Has previously received rTMS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by number of participants recruited | At consent
  Number of participants recruited will serve as a measure of study feasibility. Target enrollment is 50 participants.
Feasibility as measured by the percent of participants who complete the study | 3-month follow-up
  The percent of participants who complete the 3-month follow-up visit will serve as a measure of treatment feasibility. 80% retention will be the cut point.
Number of participants with self-reported and bioverified abstinence from smoking | End of treatment, about five weeks after beginning study
  Effectiveness of the intervention will be measured by the number of participants who self-report 7-day point prevalence at the end of treatment, and self-report is bioverified by exhaled carbon monoxide.
Number of participants with self-reported and bioverified abstinence from smoking | 3-month follow-up
  Effectiveness of the intervention will be measured by the number of participants who self-report 7-day point prevalence at the 3-month follow-up visit, and self-report is bioverified by salivary cotinine.

SECONDARY OUTCOMES:
Average number of cigarettes smoked per day in past week | End of treatment, about five weeks after beginning study
  Participants will self-report the number of cigarettes they have smoked per day in the past week.
Average number of cigarettes smoked per day in past week | 3-month follow-up
  Participants will self-report the number of cigarettes they have smoked per day in the past week.
Self-reported withdrawal symptoms | End of treatment, about five weeks after beginning study
  Participants will self-report withdrawal symptoms on the Minnesota Nicotine Withdrawal Scale. Scores on this scale range from 0 to 36, with higher scores indicating higher severity of withdrawal symptoms.
Self-reported withdrawal symptoms | 3-month follow-up
  Participants will self-report withdrawal symptoms on the Minnesota Nicotine Withdrawal Scale. Scores on this scale range from 0 to 36, with higher scores indicating higher severity of withdrawal symptoms.
Self-report of craving based on Questionnaire of Smoking Urges | End of treatment, about five weeks after beginning study
  Participants will self-report cravings for tobacco on the Questionnaire of Smoking Urges. Scores on this scale range from 0 to 60, with higher scores indicating higher smoking craving.
Self-report of craving based on Questionnaire of Smoking Urges | 3-month follow-up
  Participants will self-report cravings for tobacco on the Questionnaire of Smoking Urges. Scores on this scale range from 0 to 60, with higher scores indicating higher smoking craving.
Number of participants who report relapse to smoking | End of treatment, about five weeks after beginning study
  Measured by self-report, smoking relapse is defined as smoking 5 or more cigarettes per day for 3 consecutive days.
Number of participants who report relapse to smoking | 3-month follow-up
  Measured by self-report, smoking relapse is defined as smoking 5 or more cigarettes per day for 3 consecutive days.
Functional network connectivity changes | End of repetitive transcranial magnetic stimulation treatment, about three weeks after beginning study
  Comparison of functional network connectivity (FNC) changes between the postcentral gyrus cortical rTMS target and right posterior insula using magnetic resonance imaging before and after the rTMS course
Neuroimaging correlates to tobacco use | End of repetitive transcranial magnetic stimulation treatment, about three weeks after beginning study
  Correlation of resting state functional connectivity changes pre- vs post-rTMS course and the change in the number of cigarettes smoked in the past 24 hours
Self-report of craving based on Urge to Smoke Scale | End of treatment visit, about five weeks after beginning study
  Participants will report smoking craving using this single-item measure. Scores range from 0 to 100 with higher scores indicating higher smoking craving.
Self-report of craving based on Urge to Smoke Scale | 3-month follow-up
  Participants will report smoking craving using this single-item measure. Scores range from 0 to 100 with higher scores indicating higher smoking craving.
Self-report of craving based on Urge to Smoke Scale | End of treatment, about five weeks after beginning study
  Participants will self-report craving on the single-item Urge to Smoke Scale. Scores on this scale range from 0 to 100, with higher scores indicating higher cravings to smoke.
Self-report of craving based on Urge to Smoke Scale | 3-month follow-up
  Participants will self-report craving on the single-item Urge to Smoke Scale. Scores on this scale range from 0 to 100, with higher scores indicating higher cravings to smoke.

OTHER OUTCOMES:
Self-report posttraumatic stress disorder (PTSD) symptoms | End of treatment, about five weeks after beginning study
  Participants will self-report PTSD symptoms on the PTSD Checklist - 5. Scores on this measure range from 0 to 80, with higher scores indicating higher severity of PTSD symptoms.
Self-report posttraumatic stress disorder (PTSD) symptoms | 3-month follow-up
  Participants will self-report PTSD symptoms on the PTSD Checklist - 5. Scores on this measure range from 0 to 80, with higher scores indicating higher severity of PTSD symptoms.
Self-reported depressive symptoms | End of treatment, about five weeks after beginning study
  Participants will self-report depression symptoms on the Inventory of Depressive Symptomatology. Scores on this scale range from 0 to 90, with higher scores indicating higher depression symptom severity.
Self-reported depressive symptoms | 3-month follow-up
  Participants will self-report depression symptoms on the Beck Depression Inventory - 2. Scores on this scale range from 0 to 63, with higher scores indicating higher depression symptom severity.
Severity of baseline smoking on abstinence | End of treatment, about five weeks after beginning study
  Measured by self-report, plan to evaluate degree of baseline smoking severity (daily cigarettes) on smoking abstinence at end-of-treatment
Severity of baseline smoking on abstinence | 3-month follow-up
  Measured by self-report, plan to evaluate degree of baseline smoking severity (daily cigarettes) on smoking abstinence at 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Young, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No